CLINICAL TRIAL: NCT06629259
Title: Guanfacine for Alcohol Use Disorder (AUD): a Telehealth Approach
Brief Title: Guanfacine for Alcohol Use Disorder (AUD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Helen Fox, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 24432; R01AA031662-01 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-10-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Stress; Guanfacine; Sex Differences
MeSH Terms: conditions — Alcoholism | interventions — Guanfacine

STUDY DESIGN:
Intervention Model Description: randomized double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Guanfacine Extended Release (XR) (Experimental): Participants receive guanfacine XR, 3mg tablet orally, once per day for 12 weeks
  Interventions: Drug: Guanfacine Extended Release (XR)
- Placebo (Placebo Comparator): Participants receive guanfacine XR, placebo tablet orally, once per day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine Extended Release (XR) — 3mg tablet once daily
  Other Names: Intuniv
  Arms: Guanfacine Extended Release (XR)
Drug: Placebo — placebo tablet once daily
  Arms: Placebo

SUMMARY:
The investigators assess whether guanfacine extended release (GXR; 3mg/d) compared with placebo (PBO) will attenuate drinking and drinking-related factors in N=200 men and women with Alcohol Use Disorder (AUD) across 12-weeks.

DETAILED DESCRIPTION:
This is a study to examine the efficacy of guanfacine extended release (GXR) (3mg/d) compared with placebo (PBO) in reducing drinking in N=200 men and women with Alcohol Use Disorder (AUD). The study will be conducted across two sites for 12-weeks. Indiana University will be the primary site and Rutgers University, the secondary site. Participants at both sites will be randomized to either GXR (3mg/d) or placebo (PBO), and titrated to full dose over a three week period. After remaining at full dose for 7 weeks a two week schedule will be used to taper participants off the medication. During the study the investigators will collect brief reports throughout the day and evening of drinking severity, stress, craving, mood, arousal, anxiety, and emotion regulation at weeks 1 and 2 (baseline) and weeks 5 and 6 (steady state). Additionally, blood alcohol concentration (BAC) levels will be collected three times per day for the full 12-weeks. Daily encrypted video recordings will be used to monitor medication compliance, and participants will also take part in twice weekly remote visits to assess safety, vitals, collect urines, monitor alcohol use, and receive weekly Medical Management. It is anticipated that guanfacine will demonstrate greater efficacy in women compared to men with AUD.

ELIGIBILITY:
Inclusion Criteria:

* be assigned as a biological male or female at birth and identify as such
* meet current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM V) criteria for moderate to severe AUD
* be ≥18 years old and have a body mass index (BMI) of 18-35
* express a desire to quit alcohol as determined by the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES)
* demonstrate a positive urine for alcohol on admission to study procedures
* be able to provide informed verbal and written consent
* be able to read English and complete study evaluations
* be in good health as verified by the intake 1 physical examination

Exclusion Criteria:

* meet criteria for moderate to severe Substance Use Disorder (SUD), excluding alcohol and nicotine
* have a positive screen for substances of abuse, excluding alcohol, nicotine,
* being psychotic or otherwise severely psychiatrically disabled (including suicidal, homicidal, current mania)
* meet criteria for physiological dependence on alcohol requiring medical detoxification
* regular use of medications in the last 6 months that, in the opinion of the site physician may be contraindicated with GXR and be potentially harmful to the participant
* be pregnant or breast feeding
* be using monophasic contraceptives
* have cardiovascular disease including high blood pressure,
* be hypotensive with sitting blood pressure below 100/50 mmHG
* have bradycardia with a sitting heart rate (HR) of <60 bpm
* show EKG evidence of any clinically significant conduction abnormalities, including a Bazett's corrected QT interval (QTc) >470 msec for women and QTc>450 msec for men.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — must be assigned as a biological male or female at birth, and identify as such
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-09-07 (Estimated)

PRIMARY OUTCOMES:
Change in % number of days drinking | five times daily during weeks 1, 2, 5, 6 and twice weekly through week 12
  Self-reports of alcohol use
Change in Blood Alcohol Concentration (BAC) levels | three times per day through week 12.
  BAC levels will be collected using a remote breathalyzer application called BACtrack
Change in no. of drinks consumed following stress | five times daily during weeks 1, 2, 5, 6
  Self reports of alcohol use will be collected following stress, which will be measured using a visual analog scale (VAS) anchored from 0 (not stressed at all) to 100 (extremely stressed).
Change in alcohol craving following stress | five times daily during weeks 1, 2, 5, 6
  Self-reports of alcohol craving will be collected using a VAS anchored from 0 (Not craving at all) to 100 (Craving extremely) following self-reported stress. The VAS for stress will be anchored from 0 (not stressed at all) to 100 (extremely stressed).

SECONDARY OUTCOMES:
Change in number of drinks consumed per occasion | five times daily during weeks 1, 2, 5, 6 and twice weekly through week 12
  Self-reports of alcohol use
Change in number of binge episodes | five times daily during weeks 1, 2, 5, 6 and twice weekly through week 12
  Self-reports of alcohol use
Change in negative mood following stress | five times daily during weeks 1, 2, 5, 6
  Self-reports of negative mood will be collected using The Positive and Negative Affect Schedule (PANAS) following self-reported stress (visual analog scale; VAS). The PANAS is scored from 10-50, with a higher score representing greater negative mood. The VAS for stress will be anchored from 0 (not stressed at all) to 100 (extremely stressed).
Change in anxiety following stress | five times daily during weeks 1, 2, 5, 6
  Self-reports of anxiety will be collected using The Positive and Negative Affect Schedule (PANAS) following self-reported stress (visual analog scale; VAS). The PANAS is scored from 10-50, with a higher score representing greater anxiety. The VAS for stress will be anchored from 0 (not stressed at all) to 100 (extremely stressed).
Change in arousal following stress | five times daily during weeks 1, 2, 5, 6
  Self-reports of arousal will be collected using The Positive and Negative Affect Schedule (PANAS) following self-reported stress (visual analog scale; VAS). The PANAS is scored from 10-50, with a higher score representing greater arousal. The VAS for stress will be anchored from 0 (not stressed at all) to 100 (extremely stressed).
Change in emotion regulation following stress | five times daily during weeks 1, 2, 5, 6
  Self-reports of emotion regulation will be collected using The Difficulties in Emotion Regulation Scale (DERS) developed for ecological momentary assessment (EMA) following self-reported stress (visual analog scale; VAS). The DERS is scored from 36-180 across all items, with a higher score representing greater difficulties in regulating emotion. The VAS for stress will be anchored from 0 (not stressed at all) to 100 (extremely stressed).

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Fox, PhD, Principal Investigator — Associate Professor
Locations (2):
- United States (2):
  - The Stark Neuroscience Building (Goodman Hall), Indianapolis, Indiana
  - Rutgers School of Health Professionals, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No